CLINICAL TRIAL: NCT02773212
Title: Targeting Anhedonia in Cocaine Use Disorder - Treatment Study
Brief Title: Targeting Anhedonia in Cocaine Use Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Margaret.C.Wardle, Assistant Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018-0827
Record Dates: First submitted 2016-05-06; First posted 2016-05-16 (Estimated); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Cocaine-Related Disorders; Anhedonia
MeSH Terms: conditions — Cocaine-Related Disorders; Anhedonia | interventions — Dextroamphetamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- d-Amphetamine and Contingency Management (Experimental): Participants in this group will receive 4 weeks of treatment with 60mg of sustained release d-amphetamine with contingency management treatment for cocaine use disorder.
  Interventions: Drug: d-amphetamine; Behavioral: Contingency management
- d-Amphetamine alone (Active Comparator): Participants in this group will receive 4 weeks of treatment with 60mg of sustained release d-amphetamine but will not receive contingency management treatment for cocaine use disorder.
  Interventions: Drug: d-amphetamine
- Placebo and Contingency Management (Active Comparator): Participants in this group will receive 4 weeks of of placebo treatment, paired with contingency management treatment for cocaine use disorder.
  Interventions: Behavioral: Contingency management; Drug: Placebo (for d-amphetamine)

INTERVENTIONS:
Drug: d-amphetamine — Participants in this group will receive 60 mg of d-amphetamine daily for 4 weeks. There will be a 1 week run up dosing and a 1 week run-down medication period.
  Other Names: sustained release d-amphetamine; dexedrine
  Arms: d-Amphetamine alone; d-Amphetamine and Contingency Management
Behavioral: Contingency management — Contingency management is an established cocaine use disorder treatment in which individuals receive monetary rewards for abstinence.
  Arms: Placebo and Contingency Management; d-Amphetamine and Contingency Management
Drug: Placebo (for d-amphetamine) — 60 mg of riboflavin and cornstarch as needed.
  Arms: Placebo and Contingency Management

SUMMARY:
The purpose of this study is to examine anhedonia as a potential moderator of treatment outcomes for Cocaine Use Disorder (CUD). Specifically, this study will investigate how anhedonia affects outcomes in contingency management (CM) treatment for CUD and whether anhedonia mediates the effects of adjunctive treatment with a dopaminergic (DAergic) drug, d-amphetamine, on outcomes in CM for CUD, as well as investigate the contribution of anhedonia to overall CUD severity.

DETAILED DESCRIPTION:
Recent research suggests that anhedonia is a key neurobehavioral dysfunction in Cocaine Use Disorder (CUD) that contributes to treatment outcomes. Anhedonia, defined here as lack of interest or pleasure in non-drug rewards, is frequently found in CUD and is related to neural deficits, such as low striatal dopamine and deficient activation to non-drug rewards in mesocortical circuits. Interestingly, not all individuals in CUD have these deficits. Preliminary data suggests that the presence of self-reported anhedonia predicts worse outcome in contingency management (CM) treatment of CUD. Moreover, low baseline dopamine predicts failure to attain abstinence in CM while medications that enhance DA increase CM success rates and responsiveness to rewards.

This study specifically aims to test the contribution of anhedonia to overall CUD severity, the relationship of anhedonia to outcomes in CM treatment, and the mediating role of anhedonia in medication enhancement of CM in CUD. To accomplish these aims, individuals with CUD will be enrolled and will undergo 4 weeks of intensive CM treatment, either with or without treatment with the dopaminergic drug, d-amphetamine. A medication only group will be included to solely measure the effects of d-amphetamine. Anhedonia will be assessed using multi-modal subjective, psychophysiological and behavioral measures of reward functioning at baseline, and each week of treatment. Functional magnetic resonance imaging (fMRI) measures of reward functioning will also be taken at baseline and week 4 in a subset of participants (n = 24)

ELIGIBILITY:
Inclusion Criteria:

* be between 18 and 60 years of age
* meet Diagnostic and Statistical Manual V (DSM-5) criteria for current cocaine use disorder of at least moderate severity (≥ 4 symptoms)
* have at least 1 cocaine positive urine sample during the baseline screening period
* be in acceptable health on the basis of interview, medical history and physical exam, per the judgment of our study physician
* be able to understand the consent form and provide written informed consent
* be able to provide the names of at least 2 persons who can generally locate their whereabouts.
* if female, agree to use an acceptable method of birth control during study (surgical sterilization, approved hormonal contraceptives, barrier methods with spermicide, or intrauterine device).

Exclusion Criteria:

* current DSM-5 diagnosis for substance use disorder of least moderate severity (≥ 4 symptoms), other than cocaine, nicotine, marijuana, or alcohol
* Physical dependence on alcohol requiring medically supervised detoxification, in the judgment of the study physician
* current amphetamine use (by self-report in past 30 days or positive urine drug screen), more than 50 lifetime uses of amphetamine, or history of DSM-5 Amphetamine Use Disorder
* a current DSM-5 axis I psychiatric disorder or neurological disease or disorder requiring ongoing treatment and/or making study participation unsafe
* significant current suicidal or homicidal ideation
* medical conditions contraindicating d-amphetamine (e.g., significant cardiovascular disease, liver or kidney disease, seizure disorder, hypotension or hypertension)
* taking medications known to have effects on the central nervous system or that could cause significant drug interactions with d-amphetamine (e.g., clonidine, prazosin)
* having conditions of probation or parole requiring reports of drug use to officers of the court
* impending incarceration
* pregnant or nursing for female patients
* inability to read, write, or speak English

Additional Exclusion Criteria for the functional magnetic resonance (fMRI) Sub-Study (in addition to all listed criteria above for the Main Treatment Study):

* body mass index (BMI) >30, as this may be incompatible with the magnetic resonance scanner gantry
* any retained metals in the body, including implants and metallic substances (e.g. aneurysm clips, retained metal particles in metal workers, magnetic dental implants, ferromagnetic ocular implants, iron-based facial tattoos), as this may cause adverse effects to participants and interfere with data collection in the MR magnetic field
* inability to tolerate small, enclosed spaces (such as the magnetic resonance scanner bore)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2022-04-04 (Actual); Study Completion 2022-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret C Wardle, Ph.D., Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
All the individual participant data collected in the trial will be made available after deidentification via signed data use agreement. The study protocol and data analysis plan will also be made available.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available beginning immediately and for 3 years following the last publication from this data
Access Criteria: Data will be made available to researchers who provide a methodologically sound proposal, and to achieve the aims in the approved proposal. Proposals should be directed to mwardle@uic.edu. To gain access, data requestors will need to sign a data access agreement that will provide that the data be used solely for research and that no individuals will be identified in any manner, that data will be secured by appropriate electronic safeguards, and that once data analysis is complete, the data will be returned or destroyed. After the agreement is signed the PI will provide the necessary data to achieve proposal aims via an agreed-upon electronic method (e.g. Box Drive, university e-mail etc.)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants completed the baseline measures of anhedonia after consent but before assignment to group. Two participants were consented but not randomized - 1 due to high blood pressure at the baseline session, 1 lost to followup before completing the baseline session
Period: Overall Study
Arm/Group | d-Amphetamine and Contingency Management | d-Amphetamine Alone | Placebo and Contingency Management
Started | 21 | 15 | 19
Completed | 6 | 9 | 16
Not Completed | 15 | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | d-Amphetamine and Contingency Management | d-Amphetamine Alone | Placebo and Contingency Management | Total
Number analyzed (Participants) | 21 | 15 | 19 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.91 (7.17) | 51.87 (6.40) | 50.74 (6.11) | 51.22 (6.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 2 | 9
  Male | 16 | 13 | 17 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 3 | 8
  Not Hispanic or Latino | 18 | 13 | 16 | 47
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 2
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 16 | 12 | 16 | 44
  White | 2 | 1 | 0 | 3
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 21 | 15 | 19 | 55
Years of Education [Mean (Standard Deviation); unit: years] | 14.29 (1.59) | 13.20 (2.21) | 12.42 (1.54) | 13.34 (1.91)
Monthly Income in Dollars [Mean (Standard Deviation); unit: USD] | 1796.82 (1467.82) | 1858 (2217.13) | 1390.57 (1350.00) | 1673.18 (1650.29)
Location of Enrollment [Count of Participants; unit: Participants]
  Chicago | 14 | 4 | 8 | 26
  Houston | 7 | 11 | 11 | 29

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Were Cocaine Abstinent as Assessed by Urine Screening (Measure of Treatment Efficacy)
Description: Subjects will complete a urine drug screen each visit. Achievement of cocaine abstinence will be defined as two consecutive weeks of cocaine-negative urine samples.
Time Frame: At end of active treatment (Treatment week 4)
Measure: Count of Participants; unit: Participants
Arm/Group | d-Amphetamine and Contingency Management | d-Amphetamine Alone | Placebo and Contingency Management
Number analyzed (Participants) | 21 | 15 | 19
Participants | 3 | 3 | 6

2. Secondary Outcome: Cocaine Negative Urine Samples
Description: Subjects will complete a urine drug screen each visit (3x weekly). The Treatment Effectiveness Score is defined as the total number of cocaine negative urines across the 4 weeks of treatment (possible total of 12).
Time Frame: At end of active treatment (Treatment week 4)
Measure: Mean (Standard Deviation); unit: count of urines (range 0 - 12)
Arm/Group | d-Amphetamine and Contingency Management | d-Amphetamine Alone | Placebo and Contingency Management
Number analyzed (Participants) | 21 | 15 | 19
count of urines (range 0 - 12) | 1.76 (4.00) | 3.33 (4.25) | 5.00 (4.88)

ADVERSE EVENTS:
Time Frame: 7 weeks
Arm/Group | d-Amphetamine and Contingency Management | d-Amphetamine Alone | Placebo and Contingency Management
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/15 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/15 | 1/19
Other Adverse Events (participants affected / at risk) | 11/21 | 11/15 | 17/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | d-Amphetamine and Contingency Management (N=21) | d-Amphetamine Alone (N=15) | Placebo and Contingency Management (N=19)
Peritonsillar Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | d-Amphetamine and Contingency Management (N=21) | d-Amphetamine Alone (N=15) | Placebo and Contingency Management (N=19)
Low Energy (Psychiatric disorders) | 0 | 1 | 3
Feeling Down (Psychiatric disorders) | 1 | 1 | 2
Increased Energy (Psychiatric disorders) | 1 | 3 | 2
Anxiety (Psychiatric disorders) | 1 | 1 | 1
Problems Concentrating (Psychiatric disorders) | 1 | 0 | 0
Irritable Mood (Psychiatric disorders) | 3 | 2 | 2
Hyperactivity/Restlessness (Psychiatric disorders) | 1 | 0 | 0
Drowsy (Nervous system disorders) | 1 | 0 | 1
Change in Sleep Patterns (Nervous system disorders) | 2 | 3 | 1
Abnormal Dreams (Nervous system disorders) | 0 | 1 | 0
Headache (General disorders) | 1 | 1 | 0
Blurry Vision (Eye disorders) | 0 | 0 | 1
Joint/Muscle Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 5
Heart Racing (Cardiac disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Chills (General disorders) | 0 | 1 | 0
Increased Sweating (General disorders) | 1 | 0 | 0
Tingling Skin (Nervous system disorders) | 1 | 0 | 1
Skin Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dry Mouth (General disorders) | 0 | 1 | 1
Change in Urination (Renal and urinary disorders) | 1 | 2 | 1
Change in Appetite (General disorders) | 0 | 1 | 1
Black Stools (Gastrointestinal disorders) | 0 | 0 | 1
Change in Weight (General disorders) | 0 | 1 | 0
Numb Fingers or Toes (Nervous system disorders) | 1 | 0 | 1
High Blood Pressure (Cardiac disorders) | 6 | 9 | 14 — >140 millimeters of mercury systolic or > 90 millimeters of mercury diastolic
High Heart Rate (Cardiac disorders) | 2 | 3 | 3 — >100 beats per minute at rest

LIMITATIONS AND CAVEATS:
1. Due to recruitment issues during COVID-19 pandemic trial was terminated early (57 out of a planned 80 participants enrolled)
2. Due to complications from PI move and COVID, functional magnetic resonance imaging sub-study was never initiated.
3. During COVID-19 pandemic zygomatic muscle readings were not collected, as this would have required participants to remove masks

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-16): https://cdn.clinicaltrials.gov/large-docs/12/NCT02773212/Prot_SAP_000.pdf
  • Informed Consent Form (2024-04-18): https://cdn.clinicaltrials.gov/large-docs/12/NCT02773212/ICF_002.pdf